CLINICAL TRIAL: NCT02272972
Title: Performance Improvement Program on Imaging II
Status: Completed | Type: Observational
Sponsor: AO Clinical Investigation and Publishing Documentation (Other)
Responsible Party: Sponsor
Organization: AO Innovation Translation Center (Other)
Other Study IDs: PI program II
Record Dates: First submitted 2014-10-10; First posted 2014-10-23 (Estimated); Last update posted 2020-08-13 (Actual); Status verified 2020-08

CONDITIONS: Hip Fractures; Femoral Fractures; Fractures, Bone
Keywords: "fluoroscopy"[MeSH], "education, medical"[MeSH]
MeSH Terms: conditions — Hip Fractures; Femoral Fractures; Fractures, Bone

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Retrospective group: One x-ray image per patient is assessed by the surgeon. The surgeon undergoes an educational intervention (video/poster) and applies the achieved knowledge during the second assessment of the same image. The intervention is not administered to patients, only to an image.
- Prosp.group (Application of knowledge): No direct intervention at the patient. The surgeon applies the achieved knowledge during the performance of the fluoroscopy in the operating room. This image is assessed.
  Interventions: Other: Application of knowledge

INTERVENTIONS:
Other: Application of knowledge — Educational Intervention has been performed at the treating surgeon (video and poster). The surgeons applies the achieved knowledge when performing the intraoperative fluoroscopy in patients with pertrochanteric fractures.
  Groups: Prosp.group (Application of knowledge)

SUMMARY:
This study consists of a retrospective and a prospective part. For each part and in each of 5 clinics, one intraoperative postimplant image (lateral view) of 25 patients with pertrochanteric fractures will be assessed by 5 surgeons per clinic. There are two assessments in the retrospective part. a) before an educational intervention, b) after the educational intervention. The evaluated images at these two timepoints are identical. In the prospective part, the surgeons apply their new knowledge from the educational intervention. They perform the positioning of the patient during the intraoperative fluoroscopy and record the image according to the teaching material. One postimplant image of each patient will be used for the evaluation.

At all three timepoints of image assessment, a questionnaire with the same set of 7 criteria (Q1-Q7) for assessing the radiographs is used. The criteria refer to the content of the educational material.

DETAILED DESCRIPTION:
5 surgeons in 5 clinics will participate including a total of 125 prospective and 125 retrospective cases. This means 25+25 cases per clinic or 5+5 cases treated by each surgeon. The anonymized images of the surgeon's last 5 patients (retrospective part) and the pseudonymized images of the next 5 patients meeting the eligibility criteria (prospective part) will be assessed. Patients are eligible if they are at least 18 years old, have an AO 31-A1, A2 or A3 fracture and were treated with either a Proximal Femoral nail Antirotation (PFNA), a PFNA- II, a Dynamic Hip Screw (DHS) or a Titanium Trochanteric Fixation Nail System (TFN).

Individually, the 5 surgeons per clinic review the 25 postimplant intraoperative lateral images filed for 5 retrospective cases using a set of predefined criteria.

After this first assessment of retrospective cases, the group watches a video and a poster and has one hour of time to discuss it. The group reviews the 25 cases from the pre-education step again within a period of maximum 5 days. The data are analyzed at AO Clinical Investigation and Documentation (AOCID) and provided to the surgeons for data review meeting where they agree on areas for improvement and set target goals for the prospective series. For the whole period of the second assessment and the prospective series, the poster is placed in the area of the operating room.

After patient information/consent, eligible patients are included into the prospective part of the study and treated with either an intramedullary nail or a DHS. During the surgery, the surgeons use the newly achieved knowledge to record images.

In the next step, the 5 surgeons per clinic review individually 25 postimplant intraoperative lateral images of 5 prospective cases using the same set of predefined criteria. The data are analyzed at AOCID and review by the Imaging Working Group of AO Education.

The data are not transferred between the clinics. The main outcomes will be assessed based on the "Questionnaire for the assessment of the lateral intraoperative view of the proximal femur".

This questionnaire consists of seven questions, on image quality (Q1 and Q2; part A) and on quality of reduction and surgery (Q3 - Q7; part B). Q1 and Q2 allow only "yes/no" answers, with an option to comment on the answer "no". Q3 to Q5 are based on anatomical assessments and Q6 and Q7 ask for evaluation of the surgery. There is a "not assessable" answer option for all questions of part B.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years and older
* Diagnosis of a pertrochanteric femoral fracture (AO 31-A1, A2, A3)
* Surgical treatment with either a Proximal Femoral Nail Antirotation (PFNA), a PFNA-II, a Dynamic Hip Screw (DHS) or a Titanium Trochanteric Fixation Nail System (TFN)

For the prospective part of the study:

Informed consent obtained, i.e.:

* Ability to understand the content of the patient information/Informed Consent Form
* Willingness to allow the use of health-related data (images) according to the Clinical Investigation Plan (CIP)
* Signed and dated Ethics Committee (EC)/Institutional Review Board (IRB) approved written informed consent

Exclusion Criteria:

For the prospective part of the study: - Mentally handicapped patients or patients with dementia that are not able to understand the content patient information/Informed Consent Form

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients are eligible if they are at least 18 years old, have an AO 31-A1, A2 or A3 fracture and were treated with either a Proximal Femoral nail Antirotation (PFNA), a PFNA- II, a Dynamic Hip Screw (DHS) or a Titanium Trochanteric Fixation Nail System (TFN).
Sampling Method: Non-Probability Sample
Enrollment: 250 (Actual)
Dates: Start 2014-10; Primary Completion 2016-04 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Image quality as determined by The proportion of "yes" answers to Q1 and Q2 in the post-educational assessment II compared to the proportion of "yes" answers to Q1 and Q2 pre-educational assessment. | 6 months

SECONDARY OUTCOMES:
Interrater agreement between pre-educational and post-educational assessment of image quality (Q1-Q2) | 6 months
Proportion of images that are rated as "not assessable" (Q3-Q7) | 6 months
Proportion of "Quality of reduction and surgery" criteria with the best possible assessment (yes/optimal) (Q3-Q7) | 6 months
Interrater agreement between pre-educational and post-educational assessment of surgery's quality (Q3-Q7) | 6 months
Surgeons' experience (years and professional level) | 6 months
Surgeons practice (average number of hip surgeries per month) | 6 months
Self-assessment gap score | 6 months
  (3 questions regarding the current and the desired level of ability in fixing pertrochanteric femoral fractures, obtaining lateral intraoperative images of the proximal femur and assessing lateral intraoperative images of the proximal femur)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Rikli, MD, Principal Investigator — University Hospital, Basel, Switzerland
Locations (5):
- University of Missouri Hospital and Clinics, Columbia, Missouri, United States
- Hospital of the Medical University Graz, Graz, Austria
- University Medical Centre Ljubljana, Ljubljana, Slovenia
- Switzerland (2):
  - Cantonal Hospital Winterthur, Winterthur, Canton of Zurich
  - Municipal Hospital Triemli, Zurich, Canton of Zurich

REFERENCES:
- [Background] Heetveld MJ, Raaymakers EL, van Walsum AD, Barei DP, Steller EP. Observer assessment of femoral neck radiographs after reduction and dynamic hip screw fixation. Arch Orthop Trauma Surg. 2005 Apr;125(3):160-5. doi: 10.1007/s00402-004-0780-4. Epub 2005 Mar 2. PMID 15742193
- [Background] Karanicolas PJ, Bhandari M, Walter SD, Heels-Ansdell D, Sanders D, Schemitsch E, Guyatt GH. Interobserver reliability of classification systems to rate the quality of femoral neck fracture reduction. J Orthop Trauma. 2009 Jul;23(6):408-12. doi: 10.1097/BOT.0b013e31815ea017. PMID 19550226
- [Background] Rushton MN, Rushton VE, Worthington HV. The value of a quality improvement programme for panoramic radiography: a cluster randomised controlled trial. J Dent. 2013 Apr;41(4):328-35. doi: 10.1016/j.jdent.2012.12.009. Epub 2013 Jan 18. PMID 23337088
- [Background] Zisblatt L, Kues JR, Davis N, Willis CE. The long-term impact of a performance improvement continuing medical education intervention on osteoporosis screening. J Contin Educ Health Prof. 2013 Fall;33(4):206-14. doi: 10.1002/chp.21200. PMID 24347099
- [Background] Cannon CP, Hoekstra JW, Larson DM, Karcher RB, Mencia WA, Berry CA, Stowell SA. A report of quality improvement in the care of patients with acute coronary syndromes. Crit Pathw Cardiol. 2011 Mar;10(1):29-34. doi: 10.1097/HPC.0b013e318204eb8b. PMID 21562372
- [Background] Krettek C, Miclau T, Grun O, Schandelmaier P, Tscherne H. Intraoperative control of axes, rotation and length in femoral and tibial fractures. Technical note. Injury. 1998;29 Suppl 3:C29-39. doi: 10.1016/s0020-1383(98)95006-9. PMID 10341895